CLINICAL TRIAL: NCT02217696
Title: Neuronal Markers of Grapheme-phoneme Training Response for Prediction of Successful Reading Acquisition in Children at Familial Risk for Developmental Dyslexia
Brief Title: Prediction and Intervention in Developmental Dyslexia
Acronym: LEXI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LEXI SNF32003B_141201/1; 32003B_141201/1 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Developmental Dyslexia
Keywords: Electroencephalography (EEG); Magnetic Resonance Imaging (MRI); Multimodal Neuroimaging; Development; Prediction; Intervention
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized reading training first (Experimental): Cross-over design: group first receives the intervention
  Interventions: Other: Computerized reading training
- Waiting Control First (Experimental): Cross-over design: group first serves as waiting control
  Interventions: Other: Computerized reading training

INTERVENTIONS:
Other: Computerized reading training

SUMMARY:
The long-term goal of this study is to improve prediction of poor reading outcome at preschool age by using a combination of behavioural and neuroimaging measures and to evaluate a specific computerized training program to support children with problems during reading acquisition.

ELIGIBILITY:
Inclusion Criteria for all groups:

* Healthy, native (CH-) German speaking subjects, with an estimated non-verbal intelligence quotient (IQ) >=80, without neurological and/or psychiatric disorder (except for attention deficit hyperactivity disorder, specific learning disorders, developmental language impairments)
* Additional criteria for subgroups:
* Recruitment of preschoolers (aged 5.5-7.5 years):
* Healthy children with increased risk for developmental dyslexia in their second year at kindergarten
* Recruitment of children in first grade (aged 6.5-8.5years):
* Children showing impairments in learning to read (first/second grade).
* Adults (aged 20-40 years):
* Healthy, normal reading

Exclusion Criteria for all groups:

* MRI contraindications
* No history of premature delivery and/or maternal reports of severe prenatal, perinatal or postnatal complications.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Changes in reading and spelling performance | Participants will be tested at three times for the duration of the cross-sectional intervention, an expected average of 8 months
  Performance in normed reading and/or spelling (standardized tests) as a result of reading acquisition and training

SECONDARY OUTCOMES:
Developmental and training induced changes in functional brain activation and brain structure | Participants will be tested after an expected average of 8, 12 and 16 months
  Changes in activation/structure of core language network regions assessed by EEG and MRI during development, learning and training
Accuracy of prediction on reading performance outcome | Participants will be tested at T1 and on average 8 months later
  Accuracy of prediction on reading performance (standardized tests) using behavioural and/or neuroimaging measures.
  Neuroimaging measures: EEG and MRI (functional activation, structural measures from white and/or grey matter, temporal information from event-related potential and/or frequency analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Brem, PhD, Principal Investigator — University Clinics for Child and Adolescent Psychiatry, University of Zurich
Locations (1):
- University Clinics for Child and Adolescent Psychiatry, University of Zurich, Zurich, Switzerland